CLINICAL TRIAL: NCT00955149
Title: An Open Label Pilot Trial of Erlotinib (Tarceva) in Primary Sclerosing Cholangitis With Trisomy 7
Brief Title: Erlotinib for Chemoprevention in Trisomy 7 Positive Primary Sclerosing Cholangitis (PSC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal investigator: Gregory J. Gores, M.D., Mayo Clinic, Dept. of Gastroenterology and Hepatology
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 09-000516
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Primary Sclerosing Cholangitis; Trisomy 7; Cholangiocarcinoma; Chemoprevention
Keywords: Primary sclerosing cholangitis; Trisomy 7; Cholangiocarcinoma; Chemoprevention; Erlotinib
MeSH Terms: conditions — Cholangitis, Sclerosing; Cholangiocarcinoma | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Erlotinib (Tarceva) 25 mg by mouth once daily.
  Interventions: Drug: Erlotinib (Tarceva)
- Arm B (Experimental): Erlotinib (Tarceva) 50 mg by mouth once daily for 6 months
  Interventions: Drug: Erlotinib (Tarceva)

INTERVENTIONS:
Drug: Erlotinib (Tarceva) — Patients with PSC found to be positive for Trisomy 7 on biliary brushings will be treated with Erlotinib (Tarceva) at a dose of 25 mg or 50 mg by mouth once daily for 6 months.

SUMMARY:
Primary sclerosing cholangitis (PSC) is a chronic inflammatory condition of the bile ducts of unknown etiology. It is characterized by diffuse inflammation and stricturing of the entire biliary tree, eventually resulting in cirrhosis of the liver. Patients with PSC are at increased risk for the development of cholangiocarcinoma (CCA), a cancer arising from bile duct epithelium. This risk is estimated to be approximately 1 to 1.5% per year. It is postulated that chronic inflammatory changes in the biliary epithelium promote CCA formation. The prognosis of CCA is fatal. The only potentially curative therapy is surgical; however, only a minority of patients qualify for surgical treatment.

Several studies have demonstrated overexpression of the epidermal growth factor receptor (EGFR) in CCA cells. EGFR is a type 1 tyrosine kinase promoting cell proliferation, migration and altered cell adhesion - typical characteristics of malignant neoplasias. In CCA cells, EGFR-activation is sustained resulting in cancer progression. In human CCA samples, EGFR-expression correlates with higher histologic grade, poor prognosis, and risk of recurrence. The EGFR gene is located on the short arm of chromosome 7 (7p12). Chromosomal abnormalities of the bile duct epithelium, particularly trisomy 7 (i.e. three copies of chromosome 7) can be detected in biliary epithelial samples obtained by endoscopic retrograde cholangiopancreatography (ERCP) in PSC patients. The finding of cells with trisomy 7 has preceded the development of aneuploidy and multiple chromosomal abnormalities in a number of patients, the latter chromosomal abnormalities are characteristic of CCA. Trisomy 7 amplifies the gene for EGFR thereby presumably promoting overexpression of this growth factor receptor. In a cohort of patients with Trisomy 7 and Primary Sclerosing Cholangitis patients followed for 1 year, the rate of development of Cholangiocarcinoma was 35% (n=37, Dr. Gores, unpublished observation). Patients without cytologic abnormalities were at minimal risk for the development of CCA.

Erlotinib (Tarceva) is a human EGFR type 1 tyrosine kinase inhibitor. Tarceva received FDA approval as single agent treatment for patients with locally advanced or metastatic non-small cell lung cancer. In a randomized, double blind, placebo controlled trial of 731 patients, receiving 150 mg of Tarceva or placebo once daily, median survival was prolonged to 6.7 months from 4.7 months (p<0.001). Analysis of epidermal growth factor receptor expression (45% of total study patients) demonstrated greater survival benefit in EGFR positive patients. Tarceva in combination with Gemcitabine is also FDA approved as first line therapy in patients with locally advanced, unresectable or metastatic pancreatic cancer.

Our central hypothesis is that patients with trisomy 7 will have carcinogenic changes including EGFR overexpression. EGFR blockade will inhibit a growth/survival advantage for these premalignant clones eliminating them from the biliary epithelium. As an initial step towards testing this hypothesis, the tolerability of Tarceva in this patient population needs to be established. This study will assist in determining the safety and tolerability of Tarceva in patients with primary sclerosing cholangitis. This study will be followed by a Phase 2 randomized controlled trial of Tarceva in patients with Primary Sclerosing Cholangitis with Trisomy 7.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years of age, able to provide written informed consent.
* Diagnosis of Primary Sclerosing Cholangitis.
* Scheduled for an ERCP as part of their clinical care.
* Diagnosed with trisomy 7 on cytologic testing.
* Willingness to utilize adequate contraception (if female, evidenced by being postmenopausal for at least 6 months or using contraceptive pill; for both females and males, being surgically sterile, or using two forms of barrier contraception) from screening to at least one month after the trial.

Exclusion Criteria:

* Cholangiocarcinoma, hepatocellular carcinoma, pancreatic adenocarcinoma or other malignancy <=3 years of registration.
* Other liver disease as determined by standard clinical, serological, imaging or histological criteria.
* Secondary cause of sclerosing cholangitis (IgG cholangiopathy, autoimmune, post-surgical biliary stricture, radiation, human immunodeficiency syndrome).
* Cholestasis with a bilirubin of > 1.6 mg/dl (normal range: 0.1 - 1.0 mg/dL).
* Decompensated cirrhosis, Child-Pugh Class B or C.
* Child A cirrhosis with portal hypertension (i.e., splenomegaly, esophageal or gastric varices, or platelet count < 100,000/µl [normal range: 150 - 450 x 103/µL]).
* Transaminase (AST [norm.: 8-48 U/L], ALT [norm.: 7-55 U/L]) elevation of more than three times the upper limit of the normal range.
* Pregnancy.
* Nursing mothers.
* Uncontrolled intercurrent illness.
* Concurrent administration of CYP3A modulators, Antiepileptics, Rifampin, St. Johns wort, Ketoconazole, protonpump-inhibitors.
* Men or women unwilling to employ adequate contraception.
* Abnormalities of the cornea by history.
* Moderate diarrhea defined as defecation frequency of equal or more than 4/d for those with their colon, equal or more than 8/d for patients with a pouch, and high ostomy output with those with ostomy.
* Known interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
To examine the safety and tolerability of Tarceva (Erlotinib) in patients with primary sclerosing cholangitis and trisomy 7 on biliary cytology. | 6 months

SECONDARY OUTCOMES:
To assess among patients with primary sclerosing cholangitis and trisomy 7 the resolution of this cytologic abnormality following treatment with Tarceva (Erlotinib). | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States